CLINICAL TRIAL: NCT03351855
Title: Phase I/II and Multicenter Trial of HPV Specific Immune Lymphocytes (HPV-CTLs) in the Treatment of Human Papilloma Virus (HPV) Infection
Brief Title: HPV Specific Immune Lymphocytes (HPV-CTLs) in the Treatment of HPV
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-17020
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Human Papilloma Virus
Keywords: Human papilloma virus; Cytotoxic lymphocyte; HPV-CTL

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPV-CTLs (Experimental): Autologous or allogenic HPV specific cytotoxic lymphocytes
  Interventions: Biological: HPV-CTLs

INTERVENTIONS:
Biological: HPV-CTLs — 2 to 4 infusions, once a week, for 1x10^5~4x10^6 CTLs/kg by IV each time

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and efficacy of IV-infused autologous or allogenic HPV-CTLs.

DETAILED DESCRIPTION:
Human papilloma viruses (HPV) have been consistently implicated in causing cervical cancer especially those high-risk types (HPV 16, 18, 31, 45). Around 50-80% of women are infected by HPV within their whole lives. The current treatment of HPV-positive mainly includes drug, cryotherapy, laser, microwave, surgery and so on. Some treatments are convenient, but easy to cause pain or infection and there is still a greater risk of recurrence after treatment.

Adoptive immunotherapy with cytotoxic T lymphocytes (CTLs) reactive with specific viral antigens has proven to be effective. Here, the investigators aim to evaluate the safety and efficacy of multiple infusions of HPV specific cytotoxic T lymphocytes cells in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written, informed consent obtained prior to any study-specific procedures.
2. Evidence of HPV virus activation (viral DNA) or high risk of HPV infection.
3. Not suitable for routine treatment or invalid to antiviral drugs.
4. Patients with viral disease symptoms and confirmed by biopsy, regardless of the level of virus DNA.
5. Age less than 75 years.
6. Did not use Penicillin or β-lactam antibiotics, or the lowest dose of other antibiotics.
7. Initial hematopoietic reconstitution: neutrophils (ANC) ≥ 1,000/mm^3, platelet (PLT) ≥ 1,000/mm^3.
8. Proper renal and hepatic functions (ULN denotes "upper limit of normal range"): Creatinine ≤ 2*ULN, Bilirubin ≤ 2*ULN, SGOT/ SGPT ≤ 3*ULN.
9. If HPV-CTL is not from the patient's own, then the provider of HPV-CTL needs to meet the following criteria:

   * did not receive chemotherapy or radiotherapy within 4 weeks prior to blood collection, and did not take any steroids for the previous week, did not use Penicillin or β-lactam antibiotics, or the lowest dose of other antibiotics.
   * white blood cells ≥ 3,500 / μl, lymphocytes ≥ 750 / μl.
10. Human immunodeficiency virus (HIV) test was negative.

Exclusion Criteria:

1. Subject or the donor of BMT recipient infected with HCV (HCV antibody positive), HBV (HBsAg positive), HIV (HIV antibody positive), HTLV (HTLV antibody positive), Treponema pallidum antibody positive or TB culture positive.
2. Subject is albumin-intolerant.
3. Subject with life expectancy less than 8 weeks.
4. Subject participated in other investigational somatic cell therapies within past 30 days.
5. Subject with positive pregnancy test result.

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of HPV-CTLs in patients using CTCAE version 4.0 standard to evaluate the level of adverse events | 6 months
  Physiological parameter (measuring cytokine response, fever, symptoms)

SECONDARY OUTCOMES:
Viral load response | 6 months
  The viral load response to the CTLs infusion will be assessed by HPV specific PCR of peripheral blood.
Treatment Responses | 1 year
  Disease status is defined by the biochemical markers (measuring HPV concentration and so on) to get the outcomes such as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD).

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, PhD, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No